CLINICAL TRIAL: NCT06945952
Title: Effectiveness of the Ratio of Respiratory Rate to Diaphragm Thickening Fraction in Predicting Successful Extubation
Brief Title: Efficacy of the Ratio of Respiratory Rate to Diaphragm Thickening Fraction in Prediction of Successful Weaning
Status: Active, not recruiting | Type: Observational
Sponsor: Eman Diaa AlDin Hassan AlHassanin (Other)
Responsible Party: Sponsor-Investigator, Eman Diaa AlDin Hassan AlHassanin, principal investigator, Benha University
Organization: Benha University (Other)
Other Study IDs: md6-5-2024
Record Dates: First submitted 2025-04-08; First posted 2025-04-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Extubation Success

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: diaphragmatic ultrasonography — using diaphragmatic ultrasonography to measure diaphragmatic thickening fraction and then calculate the ratio RR/DTF

SUMMARY:
the aim of this prospective cross-sectional study is Assessment the effectiveness of the RR/DTF in predicting successful extubation . and to Compare the effectiveness of the RR/DTF with conventional parameters (RSBI, VC, PIMAX) for predicting successful extubation

All participants will undergo a SBT by using pressure support ventilation (PSV) with pressure support of 5 cm H2O and positive end-expiratory pressure (PEEP) of 5 cm water (H2O) .

The decision to start weaning, extubation or reintubation will be made based on the attending physician's discretion following local guidelines. Daily, patients will be assessed by the attending physician for weaning readiness. Investigators will be informed when the ICU attending decide to extubate.

DETAILED DESCRIPTION:
this study will be carried out on mechanically ventilated patients in medical and surgical intensive care units (ICU) at Banha University Hospitals.

Each Patient after taking an informed consent will be subjected to:

1. Full history taking including:

   Personal, present, past, family, and surgical histories of the patients will be documented. This includes collecting information about the patient's demographics, current health status, medical history, family medical history, length of mechanical ventilation(MV) until SBT, underlying disease, cause of respiratory failure and any prior surgical procedures.
2. Clinical Examination:

   A thorough clinical examination of the patients will be conducted to evaluate their general health and assess any physical signs and symptoms related to the cause of admission or other conditions. Respiratory rate will be examined as well.
3. Laboratory Investigations:

   Routine laboratory investigations will be carried out, including:

   Complete Blood Count (CBC). Coagulation studies, including Prothrombin Time (PT), Partial Thromboplastin Time (PTT), and International Normalized Ratio (INR). Renal function tests, including Urea and Creatinine levels. Liver function tests, including Serum Glutamic Oxaloacetic Transaminase (SGOT) and Serum Glutamic Pyruvic Transaminase (SGPT).
4. Procedures:

SBT

Measurements:

Exhaled tidal volume(VT), RR, RSBI, vital capacity (VC) , PIMAX, and diaphragmatic parameters will be measured in all participants at 2 h after the SBT. VT will be calculated as minute ventilation divided by RR. The RSBI will be obtained by dividing RR (breaths/min) with tidal volume (litres). Measurement of vital capacity will be performed in the upright position after measurement of minute ventilation. PIMAX will be obtained by occluding the airway at end-expiration through a unidirectional valve, a calibrated device attached to the end of an endotracheal tube. PIMAX will be the most negative pressure documented after airway occlusion when patients will be instructed to take a maximal inspiratory effort against the closed valve. Transthoracic ultrasonography will be performed at the bedside with patients in a semi-recumbent position with the head of the bed at 30- 45 degrees from three consecutive tidal breaths on each side of the hemidiaphragm, and average values will be used for analysis. The diaphragm thickening fraction (DTF) percentage will be calculated with the following formula: thickness at the end of inspiration minus thickness at the end of expiration, divided by thickness at the end of expiration, then multiplied by 100. The RR/DTF will be calculated by dividing the respiratory rate (RR) by the DTF.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Both sexes will be included.
* Patients with acute respiratory failure caused by medical or postoperative conditions who had been receiving MV for more than 48 h and tolerated 2 h spontaneous breathing trial (SBT)
* Readiness for weaning from MV (recovery from the cause of respiratory failure, hemodynamic stability in the absence of vasopressors, and no administration of neuromuscular blocking agents or sedative drugs for more than 24 h prior to enrollment).

Exclusion Criteria:

* History of neuromuscular disease or thoracic surgery.
* Pneumothorax.
* Presence of ascites.
* Tracheostomized patients.
* Poor image quality.
* Spinal cord injury.
* Arrhythmias.
* Hemodynamic instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mechanically ventilated patients in medical and surgical intensive care units
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2026-03-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
assessing the diagnostic accuracy of the respiratory rate/diaphragmatic thickening fraction that is measured by diaphragmatic ultrasound in predicting successful extubation from mechanical ventilation | 2 years
  • The diaphragm thickening fraction (DTF) will be measured by using linear probe at the anterior axillary line with the transducer placed at the intercostal space between the 7th and 8th, or 8th and 9th ribs.Then (DTF) percentage will be calculated with the following formula: thickness at the end of inspiration minus thickness at the end of expiration,divided by thickness at the end of expiration, then multiplied by 100. The RR/DTF will be calculated by dividing the respiratory rate (RR) by the DTF.

CONTACTS AND LOCATIONS:
Overall Officials: Eman AlHassanin, MS, Principal Investigator — Benha University
Locations (1):
- Benha Uneversity, Banhā, Egypt